CLINICAL TRIAL: NCT01821872
Title: A Single Centre Prospective Randomised Study to Investigate the Cerebrospinal Fluid (CSF) Pharmacokinetics of Intravenous Paracetamol in Humans
Brief Title: Paracetamol CSF Pharmacokinetics Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 7258
Record Dates: First submitted 2013-03-27; First posted 2013-04-01 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Paracetamol
Keywords: paracetamol; acetaminophen; AM404; CSF; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sampling at approx 15 minutes (Active Comparator): Plasma and CSF samples to be taken at 15 minutes post administration of intravenous paracetamol
  Interventions: Drug: Administration of paracetamol
- Sampling at approx 30 minutes (Active Comparator): Plasma and CSF samples to be taken at 30 minutes post administration of intravenous paracetamol
  Interventions: Drug: Administration of paracetamol
- Sampling at approx 120minutes (Active Comparator): Plasma and CSF samples to be taken at 120 minutes post administration of intravenous paracetamol
  Interventions: Drug: Administration of paracetamol

INTERVENTIONS:
Drug: Administration of paracetamol — Administration of 1g intravenous paracetamol
  Other Names: Perfalgan

SUMMARY:
Despite its use for decades all over the world, the exact mechanism of action of paracetamol is not fully understood and essentially involves a combination of hypotheses. It is known to have an effect via the central nervous system, and of the many mechanisms proposed, one hypothesis is that it may have indirectly activate CB1 (cannabinoid) receptors, through its novel metabolite AM404.

This study aims to elucidate cerebrospinal levels of paracetamol and to measure the concentration of its metabolites, including AM404 in CSF. This may, in turn, give us useful information on the mechanism of action of paracetamol.

DETAILED DESCRIPTION:
Patients undergoing spinal blockade for urological surgery were administered 1g paracetamol intravenously at varying intervals prior to spinal anaesthesia, at which time 5mls of cerebrospinal fluid and 10mls of blood were sampled, and analysed for concentrations of paracetamol, paracetamol glucuronide, paracetamol sulphate, and AM404, a known endocannabinoid reuptake inhibitor, and metabolite of paracetamol.

Paracetamol readily penetrates into the cerebrospinal fluid in animal studies and in children. This could account for the rapid central analgesic and antipyretic action of intravenous paracetamol however this remains to be studied in adults. AM404 has never before been identified in humans, and its presence in CSF following paracetamol supports the hypothesis of a central mechanism of action of paracetamol via AM404.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18 to 80 years
* Subjects undergoing surgery who require a spinal anaesthetic and paracetamol as part of their routine anaesthetic plan
* Subjects with an American Society of Anesthesiology score of I-III

Exclusion Criteria:

* Subjects with any contraindication to spinal anaesthesia
* Subjects with known clotting abnormalities
* Pregnant or lactating women
* Subjects with known hypersensitivity to paracetamol
* Patients with severe hepatocellular insufficiency
* Patients already taking regular doses of paracetamol
* Any subjects deemed medically unsuitable by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Measurement of AM404 in CSF | 5-211 minutes post-administration of paracetamol
  AM404 is a metabolite of paracetamol thought to be formed in the brain.

SECONDARY OUTCOMES:
Measurement of paracetamol in plasma and CSF | 5-211 minutes post administration of paracetamol
  Concentrations of paracetamol measured in plasma and CSF following intravenous paracetamol administration.
Measurement of paracetamol glucuronide and sulphate conjugates in plasma and CSF. | 5-211 minutes post administration of paracetamol
  Concentrations of glucuronide and sulphate conjugates of paracetamol measured in plasma and CSF following intravenous paracetamol administration.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Mehta, MD, Study Director — Pain and Anaesthesia Research Centre, Barts Health NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom